CLINICAL TRIAL: NCT04566822
Title: Testing the Feasibility and Preliminary Effects of a Six-week Online Program, "Calm Sleep Coaching", in Adults With Sleep Disturbance
Brief Title: Calm Sleep Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00012385
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: The participants will be blinded as to which group is receiving the intervention being assessed
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-touch intervention (Experimental): * 6 live video coaching sessions
  * Coaching/feedback is tailored to the individual and adaptive to their progress
  * Member can send the Coach messages between sessions, but the Coach will not respond until the live session
  Interventions: Behavioral: High Touch intervention
- medium-touch intervention (Experimental): * 3 live video coaching sessions
  * 2 live videos are optional (recommended for end of Weeks 3 and 5, but member can take advantage of them anytime)
  * 2-4 pre-recorded video sessions at end of the week. Pre-recorded videos provided in the absence of live sessions
  * Chat messaging between sessions with 24-48 hour response time
  Interventions: Behavioral: Medium Touch intervention
- low-touch intervention (Experimental): * 1 Live video coaching session (week 1)
  * Chat messaging with 24-48 hour response time
  Interventions: Behavioral: Low Touch intervention
- Sleep education control (Sham Comparator): * Weekly sleep education for six weeks
  * No interaction with coach
  Interventions: Behavioral: Sleep Education Control

INTERVENTIONS:
Behavioral: High Touch intervention — The Calm app is downloadable by participants onto their smartphone to access the Calm app and Calm Sleep Coaching. The Calm app is used to deliver the intervention to experimental group participants.
  Arms: High-touch intervention
Behavioral: Medium Touch intervention — The Calm app is downloadable by participants onto their smartphone to access the Calm app and Calm Sleep Coaching. The Calm app is used to deliver the intervention to experimental group participants.
  Arms: medium-touch intervention
Behavioral: Low Touch intervention — The Calm app is downloadable by participants onto their smartphone to access the Calm app and Calm Sleep Coaching. The Calm app is used to deliver the intervention to experimental group participants.
  Arms: low-touch intervention
Behavioral: Sleep Education Control — Participants in the sleep education control will not have access to a coach. Weekly sleep education will be accessible to the participant on a weekly basis. The sleep education content will be the same that is provided to the intervention participants.
  Arms: Sleep education control

SUMMARY:
The Centers for Disease Control and Prevention has identified insufficient sleep as a public health epidemic, with more than 70 million US adults experiencing insomnia each year. However, access to current evidence-based interventions for sleep disturbance (e.g., Cognitive Behavior Therapy for Insomnia [CBT-I]) is limited due to the need for specialized providers as well as monetary and logistical barriers that prevent many individuals from attending in-person treatment sessions (e.g., scheduling, transportation, childcare). Novel modes of delivery are needed to extend the benefits of these treatments to a wider range of individuals in need.

The purpose of this study is to evaluate Calm Sleep Coaching in adults with sleep disturbance (score of greater than or equal to 8 on the Insomnia Severity Index) by 1) determining the feasibility (i.e., acceptability, demand) of Calm Sleep Coaching and 2) determining the preliminary effects of Calm Sleep Coaching on primary (sleep quality) and secondary outcomes (i.e., symptoms of insomnia, mental health, well-being, resilience, and productivity). Investigators also aim to explore coaches' experiences with implementation of Calm Sleep Coaching using an investigator developed survey and assess the participants stage of change (transtheoretical model) throughout the program. Investigators hypothesize that 1) Calm Sleep Coaching will be feasible among individuals with sleep disturbance and 2) participating in the Calm Sleep Coaching program is associated with improvements in primary and secondary outcomes compared to the control group (with greater improvements observed among those participating in higher touch coaching interventions).

Investigators aim to recruit N=200 participants. Participants will be randomized into one of four groups: 1) High-touch intervention (N=50; real-time video and chat messaging, coach response via live videos), 2) medium-touch intervention (N=50; real-time video and pre-recorded video and chat messaging with response from coach), 3) low-touch intervention (N=50; chat messaging with response from coach), or 4) Sleep education control (N=50; no coaching).

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention has identified insufficient sleep as a public health epidemic, with more than 70 million US adults experiencing insomnia each year. However, access to current evidence-based interventions for sleep disturbance (e.g., Cognitive Behavior Therapy for Insomnia [CBT-I]) is limited due to the need for specialized providers as well as monetary and logistical barriers that prevent many individuals from attending in-person treatment sessions (e.g., scheduling, transportation, childcare). Novel modes of delivery are needed to extend the benefits of these treatments to a wider range of individuals in need.

For many individuals, digital intervention platforms may serve as an attractive alternative to receiving treatment and health services that are otherwise difficult to access. The Calm app is a consumer-based meditation smartphone app that is easy to use, inexpensive, and widely accessible (currently over 3.1 million paying subscribers). Recent surveys (N=12,151; N=11,210) indicate that between 76 and 89% of the Calm app subscribers were experiencing sleep difficulties when they downloaded the app, and 63-76% downloaded the Calm app specifically to improve their sleep. Given the Calm apps popularity and the need for techniques to improve sleep, leveraging the Calm apps existing platform will allow for efficient dissemination of a digital sleep intervention (i.e., Calm Sleep Coaching).

The Calm app has developed a new 6-week online sleep-coaching school (Calm Sleep Coaching) to improve the quality and quantity of sleep for individuals who complete the program. The development of Calm Sleep Coaching was informed by evidence-based techniques (e.g., CBTi, mindfulness practices, Self-Determination Theory, and Social Cognitive Theory). However, the feasibility and effectiveness of Calm Sleep Coaching has not yet been evaluated.

Therefore, the purpose of this study is to evaluate Calm Sleep Coaching in adults with sleep disturbance (score of greater than or equal to 8 on the Insomnia Severity Index) by 1) determining the feasibility (i.e., acceptability, demand) of Calm Sleep Coaching and 2) determining the preliminary effects of Calm Sleep Coaching on primary (sleep quality) and secondary outcomes (i.e., symptoms of insomnia, mental health, well-being, resilience, and productivity). Investigators also aim to explore coaches' experiences with implementation of Calm Sleep Coaching using an investigator developed survey and assess the participants stage of change (transtheoretical model) throughout the program. Investigators hypothesize that 1) Calm Sleep Coaching will be feasible among individuals with sleep disturbance and 2) participating in the Calm Sleep Coaching program is associated with improvements in primary and secondary outcomes compared to the control group (with greater improvements observed among those participating in higher touch coaching interventions).

Investigators aim to recruit N=200 participants. Participants will be randomized into one of four groups: 1) High-touch intervention (N=50; real-time video and chat messaging, coach response via live videos), 2) medium-touch intervention (N=50; real-time video and pre-recorded video and chat messaging with response from coach), 3) low-touch intervention (N=50; chat messaging with response from coach), or 4) Sleep education control (N=50; no coaching).

STUDY OBJECTIVES

Aim 1: Examine the feasibility (acceptability, demand) of the Calm Sleep Coaching six-week program in adults with sleep disturbance (N=200).

Acceptability is defined as participant satisfaction with content including perceived appropriateness and usefulness of Calm Sleep Coaching for improving sleep. Acceptability will be measured using an investigator developed satisfaction survey. H1.1: At least 70% of participants will report that overall, they were satisfied with Calm Sleep Coaching. H1.2: At least 70% of participants will perceive the components of Calm Sleep Coaching to be appropriate and useful for reducing or managing sleep disturbance.

Demand is defined as the number of sessions attended with the sleep coaches and compliance with sleep diaries. H1.3: At least 70% of participants will attend 4/6 of Calm Sleep Coaching sessions and (2) at least 70% will complete 70% of daily sleep diaries.

Aim 2: Test the preliminary effects of the Calm Sleep Coaching program on primary (sleep quality) and secondary outcomes (i.e., symptoms of insomnia, mental health, well-being, resilience, and productivity). Investigators will test associations between participation in Calm Sleep Coaching and changes in sleep disturbance (primary outcome) and symptoms related to sleep disturbance (secondary outcomes; i.e., stress, anxiety, depressive symptoms, well-being, resilience and productivity) compared to those in a sleep education control group. H2.1: Participating in 6 weeks of Calm Sleep Coaching will be associated with reductions in sleep disturbance. H2.2: Participating in 6 weeks of Calm Sleep Coaching will be associated with improvement in symptoms related to sleep disturbance.

Aim 3 (exploratory): Assess coaches experiences with implementation of Calm Sleep Coaching via investigator developed survey. Questions asked will assess general experiences, challenges, usability, content, and recommendations for change.

Aim 4 (exploratory): Assess the participants stage of change (transtheoretical model) throughout the program.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Own a smartphone
* Reside in the US or a US territory
* Only English speakers
* Score of greater than or equal to 8 on the Insomnia Severity Index
* Willing to download the Calm app to their smartphone
* Willing to be randomized

Exclusion Criteria:

• Greater than or equal to 60 minutes/month of meditation for the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Sleep Disturbance | Change from baseline to post-intervention (week 6)
  Sleep Disturbance will be measured with the Insomnia Severity Index. Scores range from 0-28 with higher score indicates more severe insomnia.

SECONDARY OUTCOMES:
Sleep Quality: Pittsburgh Sleep Diaries | Change from baseline to post-intervention (week 6)
  Sleep Quality will be measured using the Pittsburgh Sleep Diaries. Scores range from 0-8 with higher scores indicating greater sleep quality.
Stress | Change from baseline to post-intervention (week 6)
  Stress will be measured using the Perceived Stress Scale. Scores on the PSS-10 range from 0-40 with greater scores indicating greater stress.
Depression | Change from baseline to post-intervention (week 6)
  Depression will be measured using the Patient Health Questionnaire Depression Scale-8. Score on the PHQ-8 range from 0-24 with higher scores indicating greater depressive symptoms.
Anxiety | Change from baseline to post-intervention (week 6)
  Anxiety will be measured using the General Anxiety Disorder-7. Scores on the GAD-7 range from 0-21 with higher scores indicating greater anxiety.
Well-being | Change from baseline to post-intervention (week 6)
  Well-being will be measured using the World Health Organization-Five Well-Being Index. Scores on the WHO-5 range from 0-25 with higher scores indicating greater sense of well-being.
Resilience | Change from baseline to post-intervention (week 6)
  Resilience will be measured using the Connor-Davis Brief Resilience Scale. Scores on the CD-RISC-10 range from 0-40 with higher scores indicating greater resilience.
Productivity | Change from baseline to post-intervention (week 6)
  Productivity will be measured using the Work Productivity and Activity Impairment Questionnaire. Scores on the WPAI:GH are provided as a percentage with higher numbers indicating greater impairment and less productivity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No